CLINICAL TRIAL: NCT03213054
Title: A Phase 1 Study to Evaluate the Safety of OBP-301, Telomelysin in Combination With Radiation Therapy in Patients With Esophageal Cancer Not Applicable for Standard Therapy
Brief Title: A Study of OBP-301 With Radiation Therapy in Patients With Esophageal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oncolys BioPharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TL04001
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer; OBP-301; radiation; Telomelysin; radiotherapy; oncolytic; virotherapy; loco regional
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- OBP-301 + Radiation (Experimental): OBP-301 administration on the Day 1, Day 18 and Day 32 with standard course of radiation(total 60 Gy) for 6 weeks.
  Interventions: Biological: OBP-301; Radiation: Radiation

INTERVENTIONS:
Biological: OBP-301 — OBP-301 administration on the Day 1, Day 18 and Day 32
Radiation: Radiation — Standard radiation therapy for esophageal cancer patient. total 60 Gy for 6 weeks

SUMMARY:
This is a phase 1 study to evaluate safety and tolerability of Telomelysin (OBP-301) in combination with radiation therapy in patient with esophageal cancer who are not applicable to standard therapy.

DETAILED DESCRIPTION:
After screening, patients will undergo a combination therapy of OBP-301 with radiation therapy for 6 weeks. At Day 1, Day 18 and Day 32, OBP-301 is directly injected to the location of the lesion. From Day 4, patients receive radiation therapy. Patients will be automatically entered follow-up period for 12 weeks to be observed tolerance and safety.

This study is designated as standard 3 + 3 dose escalation study. The first 3 patients will be evaluated with low-dose of OBP-301 and then the study move onto the high-dose cohort of OBP-301. When the DLT (Dose Limiting Toxicity) is observed, 3 more patients will be enrolled in the dose level.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients who have primary tumor or metastatic lesion of histologically or cytologically diagnosed with esophageal carcinoma.
2. Patients are feasible for injection of OBP-301 into target legion
3. Patients aged in 20 to 89 years.
4. Patients with ECOG Performance Status Score ≤ 2.
5. Patient who have life expectancy longer than 12 weeks.
6. Patients who are not applicable to standard therapy.
7. Patients who have adequate organ function.

Key Exclusion Criteria:

1. Patients who have an active, treatment-required concomitant malignancy.
2. Patients who had been enrolled within 4 weeks to other clinical trials of unapproved drugs.
3. Patients who have had chemotherapy within 4 weeks.
4. Patients who have treatment history of cancer immunotherapy.
5. Patients who had radiotherapy to treatment targeted lesion.
6. Patients who have active infection which required systemic treatment.
7. Patients who are scored III or IV by NYHA (New York Heart Association).
8. Patients who are judged as inappropriate to this trial by investigator(s).

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-07-07 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicity | 18 weeks
  Occurrence of Dose Limiting Toxicity for study period to see safety and tolerability of OBP-301 combined with radiation therapy
Incidence rate of adverse event | 18 weeks
  Incidence rate of adverse event for study period to see safety and tolerability of OBP-301 combined with radiation therapy

SECONDARY OUTCOMES:
Tumor response in the treatment objected lesion | 18 weeks
  Tumor response in the treatment objected lesion within 18 weeks from the start of treatment.
Tumor response | 18 weeks
  Tumor response as the best overall response of the record within 18 weeks from the start of treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Research site, Kashima-shi, Chiba
  - Research site, Kita, Okayama-ken

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Oncolys BioPharma Homepage — http://www.oncolys.com/